CLINICAL TRIAL: NCT06810154
Title: Multi-strain Probiotics to Prevent Necrotizing Enterocolitis in Very Preterm Infants: a Stepped-Wedge Cluster Randomized Trial
Brief Title: Multi-strain Probiotics to Prevent Necrotizing Enterocolitis in Very Preterm Infants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Belal Alshaikh, Principle investigator, University of Calgary
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: U of Calgary REB24-1960
Record Dates: First submitted 2025-01-20; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Necrotizing Enterocolitis (NEC)
Keywords: Probiotics; Necrotizing enteroclitis; preterm infants
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: A Stepped-Wedge Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Infants will not receive any probiotics.
- Multi-strain probiotics (Experimental): Infants will be started on probiotics (Bifidobacterium and Lacticaseibacillus) within 24 hours of commencing enteral feeds.
  Interventions: Biological: Multi-strain probiotics

INTERVENTIONS:
Biological: Multi-strain probiotics — Infants will be started on probiotics (Bifidobacterium and Lacticaseibacillus) with enetral feed.
  Arms: Multi-strain probiotics

SUMMARY:
The goal of this clinical trial is to evaluate whether multi-strain probiotics of lactobacillus and bifidobacterium can prevent necrotizing enterocolitis (NEC) in preterm infants born at less than 32 weeks of gestation. The main questions it aims to answer are:

* Does the use of a multi-strain probiotic combination reduce the incidence of NEC in preterm infants?
* Are there any adverse effects associated with the administration of this probiotic combination?

DETAILED DESCRIPTION:
Researchers will compare outcomes between two phases:

Control Phase: No probiotics will be administered, and outcomes will be recorded to establish baseline NEC rates.

Intervention Phase: Participants will receive a daily multi-strain probiotic combination (0.5 g sachet) starting within 24 hours of enteral feeding initiation.

Participants will be:

* Preterm infants born at <32 weeks' gestation and <1500 g birth weight.

The study uses a stepped-wedge cluster randomized trial (SW-CRT) design, where neonatal intensive care units (NICUs) transition from the control phase to the intervention phase at pre-specified intervals. Individual consent will be obtained for probiotic administration and data collection during the intervention phase, and data collection-only consent will be sought during the control phase.

This trial is designed to provide high-quality evidence on the efficacy and safety of probiotics in preventing NEC in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between <32 0/7 weeks gestation.

Exclusion Criteria:

* Major congenital or chromosomal abnormalities
* Conditions affecting gastrointestinal systems that prohibit infants from starting on feed in the first 72 hours after birth.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2170 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of necrotizing enterocolitis (NEC | From date of randomization until the date of 34 weeks corrected gestational age or or date of death from any cause, whichever came first
  NEC defined in CNN according to modified Bell's criteria.

SECONDARY OUTCOMES:
Survival | From date of randomization until the date of 34 weeks corrected gestational age
Late-onset sepsis | From date of randomization until the date of 34 weeks corrected gestational age or or date of death from any cause, whichever came first
  Culture proven late onset sepsis
Growth anthropometrics at 36 weeks corrected gestation | at 36 weeks corrected age or discharge from level III NICU whichever occure first.
  Z scores of weight and head circumference
Time to achieve full enteral feed | From date of randomization until the date of 34 weeks corrected gestational age or or date of death from any cause, whichever came first
  Defined by reaching 140 mL/kg/day sustained for three consecutive days

OTHER OUTCOMES:
Probiotic sepsis | birth to discharge from level III NICU or 34 weeks corrected age whichever comes first
  Culture proven sepsis by one of the probiotics products

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Children's and Women's health of Britch Columbia, Vancouver, British Columbia
  - IWK, Halifax

IPD SHARING:
Plan to Share IPD: Undecided